CLINICAL TRIAL: NCT01974440
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of the Bruton's Tyrosine Kinase Inhibitor, PCI-32765 (Ibrutinib), in Combination With Either Bendamustine and Rituximab (BR) or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Subjects With Previously Treated Indolent Non-Hodgkin Lymphoma (iNHL)
Brief Title: A Study of PCI-32765 (Ibrutinib) in Combination With Either Bendamustine and Rituximab or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Participants With Previously Treated Indolent Non-Hodgkin Lymphoma
Acronym: SELENE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR102786; PCI-32765FLR3001 (Other: Janssen Research & Development, LLC); 2013-003093-27 (EudraCT Number)
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Results first posted 2023-04-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma
Keywords: Lymphoma; Follicular lymphoma; Marginal zone lymphoma; Indolent Non-Hodgkin lymphoma; PCI-32765; Ibrutinib; Bendamustine; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; R-CHOP
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Bendamustine Hydrochloride; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; ibrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Placebo Comparator): Treatment Arm A = background immune-chemotherapy (bendamustine and rituximab [BR] or rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone [R-CHOP]) for 6 cycles + placebo.
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Placebo
- Treatment Arm B (Experimental): Treatment Arm B = background immune-chemotherapy (BR or R-CHOP) for 6 cycles + PCI-32765 (Ibrutinib).
  Interventions: Drug: Bendamustine; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: PCI-32765 (Ibrutinib)

INTERVENTIONS:
Drug: Bendamustine — 90 milligram per meter square (mg/m^2) administered intravenously on Days 1 to 2 of Cycles 1 to 6.
Drug: Rituximab — 375 mg/m^2 administered intravenously on Day 1 of Cycles 1 to 6.
Drug: Cyclophosphamide — 750 mg/m^2 administered intravenously on Day 1 of Cycles 1 to 6.
Drug: Doxorubicin — 50 mg/m^2 administered intravenously on Day 1 of Cycles 1 to 6.
Drug: Vincristine — 1.4 mg/m^2 (maximum total 2 mg) administered intravenously on Day 1 of Cycles 1 to 6.
Drug: Prednisone — 100 mg administered orally on Days 1 to 5 of Cycles 1 to 6.
Drug: PCI-32765 (Ibrutinib) — 560 mg (4*140 mg) capsules administered orally once daily, continuously starting on Cycle 1, Day 1.
  Arms: Treatment Arm B
Drug: Placebo — Placebo (4 capsules) matched to ibrutinib administered orally once daily, continuously starting on Cycle 1, Day 1.
  Arms: Treatment Arm A

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PCI-32765 (ibrutinib) administered in combination with either bendamustine and rituximab (BR) or rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in adult participants with previously treated indolent Non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a randomized (individuals assigned to study treatment by chance), double-blind (individuals and study personnel will not know the identity of study treatments), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study in approximately 400 adult participants with follicular lymphoma or marginal zone lymphoma. The study will include the following phases: Screening, Treatment, and a Post-treatment Follow-up. Eligible participants will be randomly assigned in a 1:1 ratio to either treatment Arm A (background immune-chemotherapy + placebo) or treatment Arm B (background immune-chemotherapy + 560 milligram [mg] of ibrutinib). All participants will receive 6 cycles of background immune-chemotherapy with either BR or R-CHOP in combination with either placebo (Arm A) or ibrutinib (Arm B). Selection of background immune-chemotherapy will be based on prior treatment history and cardiac function. After completion of background immune-chemotherapy, study drug (ibrutinib or placebo) will continue until disease progression, unacceptable toxicity, or study end, whichever comes first. Assessment of tumor response and progression will be conducted in accordance with the Revised Response Criteria for Malignant Lymphoma. Serial pharmacokinetic (study of what a drug does to the body) blood samples will be collected. Safety will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of B-cell indolent Non-Hodgkin lymphoma with histological subtype limited to follicular lymphoma or marginal zone lymphoma, at initial diagnosis and without evidence of pathological transformation or clinical signs suggesting transformation
* At least 1 prior treatment with a CD20 antibody combination chemo-immunotherapy regimen
* Disease that has relapsed or was refractory after prior chemo-immunotherapy
* At least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma 2007
* Eastern Cooperative Oncology Group performance status grade 0 or 1
* Laboratory values within protocol-defined parameters
* Agrees to protocol-defined use of effective contraception
* Men must agree not to donate sperm during and after the study for 6 months after the last dose of bendamustine, 12 months after the last dose of rituximab, or 3 months after the last dose of study medication, whichever is later
* Women of childbearing potential must have a negative serum or urine pregnancy test at Screening

Exclusion Criteria:

* Prior treatment according to protocol-defined criteria
* Unable to receive background chemotherapy based on prior treatment history and cardiac function
* Known central nervous system lymphoma
* Diagnosed or treated for malignancy other than indolent Non-Hodgkin lymphoma
* History of stroke or intracranial hemorrhage within 6 months prior to randomization
* Requires anticoagulation with warfarin or equivalent Vitamin K antagonists
* Requires treatment with strong CYP3A inhibitors
* Clinically significant cardiovascular disease
* Known history of human immunodeficiency virus or active hepatitis C virus (HCV; ribonucleic acid [RNA] polymerase chain reaction [PCR]-positive) or active hepatitis B virus (HBV; DNA PCR-positive) infection or any uncontrolled active systemic infection requiring intravenous antibiotics
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the participant's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (135):
- United States (32):
  - Gilbert, Arizona
  - Campbell, California
  - Duarte, California
  - La Jolla, California
  - Los Angeles, California
  - Orange, California
  - Ocala, Florida
  - Chicago, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Westwood, Kansas
  - Lexington, Kentucky
  - Lafayette, Louisiana
  - Scarborough, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Battle Creek, Michigan
  - Detroit, Michigan
  - Saint Louis Park, Minnesota
  - Denville, New Jersey
  - New York, New York
  - Hickory, North Carolina
  - Pinehurst, North Carolina
  - Bend, Oregon
  - Pittsburgh, Pennsylvania
  - Sioux Falls, South Dakota
  - Houston, Texas
  - Lubbock, Texas
  - Spokane, Washington
  - Green Bay, Wisconsin
- Argentina (6):
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Córdoba
  - La Capital
  - Mendoza
  - Santa Fe
- Australia (6):
  - Adelaide
  - Fitzroy
  - Heidelberg
  - South Brisbane
  - Wahroonga
  - Westmead
- Belgium (6):
  - Anderlecht
  - Edegem
  - Ghent
  - Leuven
  - Namur
  - Wilrijk
- Brazil (4):
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - São Paulo
- China (8):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Harbin
  - Nanjing
  - Shanghai
  - Tianjin
- France (5):
  - Nice
  - Paris
  - Pessac
  - Pierre-Bénite
  - Rennes
- Germany (8):
  - Berlin
  - Giessen
  - Göttingen
  - Ludwigshafen
  - Magdeburg
  - Mainz
  - München
  - Wiesbaden
- Israel (7):
  - Hadera
  - Haifa
  - Jerusalem
  - Nahariya
  - Netanya
  - Petah Tikva
  - Ramat Gan
- Japan (10):
  - Chūōku
  - Hiroshima
  - Isehara
  - Kobe
  - Nagoya
  - Osaka Sayama Shi
  - Sapporo
  - Sendai
  - Suita-shi
  - Tokyo
- Poland (3):
  - Gdynia
  - Olsztyn
  - Warsaw
- Puerto Rico (3):
  - Bayamón
  - Ponce
  - San Juan
- Russia (9):
  - Krasnodar
  - Moscow
  - Nizny Novgorod
  - Petrozavodsk
  - Pyatigorsk
  - Rostov-on-Don
  - Saint Petersburg
  - Syktyvkar
  - Volgograd
- South Korea (2):
  - Jeollanam-do
  - Seoul
- Spain (4):
  - Barcelona
  - Madrid
  - Pozuelo de Alarcón
  - Salamanca
- Sweden (4):
  - Gothenburg
  - Linköping
  - Luleå
  - Uppsala
- Turkey (Türkiye) (5):
  - Ankara
  - Antalya
  - Istanbul
  - Izmir
  - Kayseri
- Ukraine (6):
  - Cherkasy
  - Ivano-Frankivsk
  - Khmelnitskiy
  - Kiev
  - Lviv
  - Uzhhorod
- United Kingdom (7):
  - Glasgow
  - London
  - Newcastle upon Tyne
  - Plymouth
  - Portsmouth
  - Sutton
  - Swansea

REFERENCES:
- [Derived] Nastoupil LJ, Hess G, Pavlovsky MA, Danielewicz I, Freeman J, Garcia-Sancho AM, Glazunova V, Grigg A, Hou JZ, Janssens A, Kim SJ, Masliak Z, McKay P, Merli F, Munakata W, Nagai H, Ozcan M, Preis M, Wang T, Rowe M, Tamegnon M, Qin R, Henninger T, Curtis M, Caces DB, Thieblemont C, Salles G. Phase 3 SELENE study: ibrutinib plus BR/R-CHOP in previously treated patients with follicular or marginal zone lymphoma. Blood Adv. 2023 Nov 28;7(22):7141-7150. doi: 10.1182/bloodadvances.2023010298. PMID 37722354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were stratified by background chemotherapy treatment (bendamustine and rituximab [BR] or combination or rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone [R-CHOP]), refractory versus relapsed disease, Indolent non-Hodgkin lymphoma histology, and number of prior lines of therapy.
Pre-assignment Details: Placebo+CIT arm participants discontinued the study treatment post the primary analysis but were assessed for the safety till the end of the study. No further efficacy analyses were done after the primary analysis.
Groups:
- Placebo + Chemoimmunotherapy (CIT): Participants received 4 capsules of placebo matching to ibrutinib orally once daily continuously starting on Cycle 1, Day 1 until disease progression, or unacceptable toxicity, or study end, whichever occurred first. All participants also received a background therapy for maximum of 6 cycles (each cycle = 21 days) either with BR: bendamustine hydrochloride 90 milligrams per meter square (mg/m^2) intravenously (IV) on Days 1 and 2 of each cycle and rituximab 375 mg/m^2 IV on Day 1 of each cycle; or background therapy with R-CHOP: rituximab 375 mg/m^2 IV on Day 1, cyclophosphamide 750 mg/m^2 IV on Day 1, doxorubicin 50 mg/m^2 IV on Day 1, vincristine 1.4 mg/m^2 IV (maximum total 2 mg) on Day 1, and prednisone 100 mg orally on Days 1 to 5 until disease progression or unacceptable toxicity. After treatment unblinding at the time of the primary analysis, participants randomized to arm "Placebo + CIT" discontinued placebo treatment.
- Ibrutinib + CIT: Participants received ibrutinib 560 mg capsules (4 capsules of 140 mg) orally once daily continuously starting on Cycle 1, Day 1 until disease progression, or unacceptable toxicity, or study end, whichever occurred first. All participants also received a background therapy for maximum of 6 cycles (each cycle = 21 days) either with BR: bendamustine hydrochloride 90 mg/m^2 IV on Days 1 and 2 of each cycle and rituximab 375 mg/m^2 IV on Day 1 of each cycle; or background therapy with R-CHOP: rituximab 375 mg/m^2 IV on Day 1, cyclophosphamide 750 mg/m^2 IV on Day 1, doxorubicin 50 mg/m^2 IV on Day 1, vincristine 1.4 mg/m^2 IV (maximum total 2 mg) on Day 1, and prednisone 100 mg orally on Days 1 to 5 until disease progression or unacceptable toxicity. After treatment unblinding at the time of the primary analysis, participants randomized to arm "Ibrutinib + CIT" continued/stopped treatment with ibrutinib at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Started | 201 | 202
Safety Analysis Set | 199 | 201
Participants With Marginal Zone Lymphoma (MZL) | 28 | 28
Participants With Follicular Lymphoma (FL) | 173 | 174
Completed | 61 | 65
Not Completed | 140 | 137
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 24 | 20
Not completed — Sponsor decision | 109 | 110

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT | Total
Number analyzed (Participants) | 201 | 202 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (12.7) | 58.9 (11.86) | 58.8 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 89 | 191
  Male | 99 | 113 | 212
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 16 | 30
  Not Hispanic or Latino | 173 | 178 | 351
  Unknown or Not Reported | 14 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 59 | 68 | 127
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 135 | 126 | 261
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 2 | 8 | 10
  AUSTRALIA | 21 | 16 | 37
  BELGIUM | 4 | 9 | 13
  BRAZIL | 1 | 2 | 3
  CHINA | 31 | 26 | 57
  FRANCE | 13 | 8 | 21
  GERMANY | 5 | 8 | 13
  ISRAEL | 16 | 17 | 33
  ITALY | 6 | 5 | 11
  JAPAN | 15 | 27 | 42
  POLAND | 4 | 4 | 8
  RUSSIAN FEDERATION | 11 | 9 | 20
  SOUTH KOREA | 12 | 14 | 26
  SPAIN | 13 | 7 | 20
  SWEDEN | 1 | 0 | 1
  TURKEY | 11 | 9 | 20
  UKRAINE | 6 | 2 | 8
  UNITED KINGDOM | 10 | 10 | 20
  UNITED STATES | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis: Progression Free Survival (PFS): Stratified Analysis
Description: PFS was defined as duration (in months) from the date of randomization to the date of disease progression or relapse from complete response (CR) or death, whichever was first reported. PFS was assessed by the investigator based on the 2007 Revised Response Criteria for Malignant Lymphoma. Disease progression was defined as any new lesion or increase by greater than or equal to (>=) 50 percent (%) of previously involved sites from nadir disease progression criteria: Appearance of new nodal lesion 1.5 centimeters (cm) in any axis, 50% increase in sum of product of diameters (SPD) of greater than (>) 1 node or 50% increase in longest diameter of previously identified node 1 cm in short axis. Participants who were progression-free and alive or had unknown status were censored at the last tumor assessment. Kaplan-Meier method was used for the analysis. Stratification factors were used for the analysis.
Time Frame: Up to 8 years
Population: Intent-to-treat (ITT) population included all randomized participants who were enrolled with follicular lymphoma (FL) or marginal zone lymphoma (MZL) and were analyzed according to the treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 201 | 202
months | 23.75 [20.11 to 31.18] | 40.51 [32.62 to 52.80]
Statistical Analysis 1: Comparison: Placebo + Chemoimmunotherapy (CIT) vs Ibrutinib + CIT; Test type: Superiority; p = 0.0922, Log Rank; Hazard Ratio (HR) = 0.806, 95% CI 2-sided [0.626 to 1.037]

2. Primary Outcome: Supplementary Analysis: Progression Free Survival: Unstratified Analysis - Participants With Marginal Zone Lymphoma (MZL)
Description: PFS in MZL participants was defined as duration (in months) from the date of randomization to the date of disease progression or relapse from CR or death, whichever was first reported. PFS was assessed by the investigator based on the 2007 Revised Response Criteria for Malignant Lymphoma. Disease progression was defined as any new lesion or increase by >=50% of previously involved sites from nadir disease progression criteria: Appearance of new nodal lesion 1.5 cm in any axis, 50% increase in SPD of >1 node or 50% increase in longest diameter of previously identified node 1 cm in short axis. Participants who were progression-free and alive or had unknown status were censored at the last tumor assessment. Kaplan-Meier method was used for the analysis. For this outcome measure, unstratified analysis was performed on participants with MZL.
Time Frame: Up to 8 years
Population: All randomized participants who were enrolled with MZL and were analyzed according to the treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 28 | 28
months | 91.63 [9.23 to NA] — "NA" represents that upper limit were not calculated due to insufficient number of participants with events | NA [49.25 to NA] — "NA" represents that median and upper limit were not calculated due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Placebo + Chemoimmunotherapy (CIT) vs Ibrutinib + CIT; Test type: Superiority; p = 0.4505, Log Rank; Hazard Ratio (HR) = 0.725, 95% CI 2-sided [0.312 to 1.682]

3. Secondary Outcome: Primary Analysis: Overall Survival (OS): Stratified Analysis
Description: OS was defined as the interval (in months) between the date of randomization and the date of the participant's death due to any cause. Kaplan-Meier method was used for the analysis. Stratification factors were used for the analysis.
Time Frame: Up to 8 years
Population: ITT population included all randomized participants who were enrolled with FL or MZL and were analyzed according to the treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 201 | 202
months | NA [94.19 to NA] — "NA" represents that median and lower limit of 95% confidence interval (CI) were not calculated due to insufficient number of participants with events. | NA [NA to NA] — "NA" represents that median and 95% CI were not calculated due to insufficient number of participants with events.

4. Secondary Outcome: Supplementary Analysis: Overall Survival: Unstratified Analysis - Participants With MZL
Description: OS in MZL participants was defined as the interval (in months) between the date of randomization and the date of the participant's death due to any cause. Kaplan-Meier method was used for the analysis. For this outcome measure, unstratified analysis was performed on participants with MZL.
Time Frame: Up to 8 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 28 | 28
months | NA [75.86 to NA] — "NA" represents that median and lower limit of 95% CI were not calculated due to insufficient number of participants with events. | NA [NA to NA] — "NA" represents that median and 95% CI were not calculated due to insufficient number of participants with events.

5. Secondary Outcome: Primary Analysis: Complete Response Rate (CRR): Stratified Analysis
Description: CRR was defined as the percentage of participants who achieved a complete response (CR); (based on investigator assessment) on or prior to the initiation of subsequent antilymphoma therapy. Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if positron emission tomography (PET) negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy and no new sites of disease detected during assessment. Kaplan-Meier method was used for the analysis. Stratification factors were used for the analysis.
Time Frame: Up to 8 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 201 | 202
percentage of participants | 50.2 | 55

6. Secondary Outcome: Supplementary Analysis: Complete Response Rate: Unstratified Analysis - Participants With MZL
Description: CRR in MZL participants was defined as the percentage of participants who achieved a CR (based on investigator assessment) on or prior to the initiation of subsequent antilymphoma therapy. Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy and no new sites of disease detected during assessment. Kaplan-Meier method was used for the analysis. For this outcome measure, unstratified analysis was performed on participants with MZL.
Time Frame: Up to 8 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 28 | 28
percentage of participants | 60.7 | 64.3

7. Secondary Outcome: Primary Analysis: Overall Response Rate (ORR): Stratified Analysis
Description: ORR was defined as the percentage of participants who achieved a CR or partial response (PR). Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy and no new sites of disease detected during assessment. Criteria for PR: >=50% decrease in sum of the diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. Kaplan-Meier method was used for the analysis. Stratification factors were used for the analysis.
Time Frame: Up to 8 years
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 201 | 202
percentage of participants | 90.5 | 91.6

8. Secondary Outcome: Supplementary Analysis: Overall Response Rate: Unstratified Analysis - Participants With MZL
Description: ORR in MZL participants was defined as the percentage of participants who achieved a CR or PR. Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy and no new sites of disease detected during assessment. Criteria for PR: >=50% decrease in sum of the diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. Kaplan-Meier method was used for the analysis. For this outcome measure, unstratified analysis was performed on participants with MZL.
Time Frame: Up to 8 years
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 28 | 28
percentage of participants | 82.1 | 89.3

9. Secondary Outcome: Primary Analysis: Duration of Response (DOR): Stratified Analysis
Description: DOR was defined as the interval (in months) between the date of initial documentation of response (CR or PR) and the date of first documented evidence of progressive disease (or relapse for participants who experienced CR during the study) or death, whichever occurred first. Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy and no new sites of disease detected during assessment. Criteria for PR: >=50% decrease in sum of the diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. Kaplan-Meier method was used for the analysis. Stratification factors were used for the analysis.
Time Frame: Up to 8 years
Population: ITT population included all randomized participants who were enrolled with FL or MZL and were analyzed according to the treatment to which they were randomized. Participants who achieved a PR or better were included in the analysis of duration of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 182 | 185
months | 21.68 [17.61 to 32.36] | 44.32 [32.89 to 60.02]

10. Secondary Outcome: Supplementary Analysis: Duration of Response: Unstratified Analysis - Participants With MZL
Description: DOR in MZL participants was defined as the interval (in months) between the date of initial documentation of response (CR or PR) and the date of first documented evidence of progressive disease (or relapse for participants who experienced CR during the study) or death, whichever occurred first. Criteria for CR: disappearance of all evidence of disease; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy and no new sites of disease detected during assessment. Criteria for PR: >=50% decrease in sum of the diameter of all target lesions compared with baseline, in absence of new lesions or unequivocal progression of non-target lesions. Kaplan-Meier method was used for the analysis. For this outcome measure, unstratified analysis was performed on participants with MZL.
Time Frame: Up to 8 years
Population: All randomized participants who were enrolled with MZL and were analyzed according to the treatment to which they were randomized. Participants who achieved a PR or better were included in the analysis of duration of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 23 | 25
months | 89.17 [42.48 to NA] — "NA" represents that upper limit of 95% CI was not calculated due to insufficient number of participants with events. | NA [73.23 to NA] — "NA" represents that median and upper limit of 95% CI were not calculated due to insufficient number of participants with events.

11. Secondary Outcome: Primary Analysis: Time to Worsening (TTW) in the Lymphoma (Lym) Subscale of the Functional Assessment of Cancer Therapy - Lymphoma Subscale (FACT-LymS) Questionnaire
Description: Time-to-worsening in the Lymphoma subscale of the FACT-Lym was defined as the time (in months) from the date of randomization to the start date of the worsening of participant symptoms. Worsening was defined by a 5-point decrease from baseline in participant symptoms. FACT-Lym Lymphoma subscale contains 15 questions, scores from 0 to 4 for each question (0 = not at all, 1 = a little bit, 2 = some what, 3 = quite a bit and 4 = very much, where the higher score indicated worse condition). Lymphoma subscale score is the total of reverse scores, range 0 to 60. Higher scores indicate a better quality of life.
Time Frame: Up to 8 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 201 | 202
months | 37.03 [24.21 to 48.33] | 24.84 [14.95 to 31.28]

12. Secondary Outcome: Supplementary Analysis: Time to Worsening (TTW) in the Lymphoma (Lym) Subscale of the Functional Assessment of Cancer Therapy - Lymphoma Subscale (FACT-LymS) Questionnaire: Participants With MZL
Description: TTW in MZL participants in the Lymphoma subscale of the FACT-Lym was defined as the time (in months) from the date of randomization to the start date of the worsening of participant symptoms. Worsening was defined by a 5-point decrease from baseline in participant symptoms. FACT-Lym Lymphoma subscale contains 15 questions, scores from 0 to 4 for each question (0 = not at all, 1 = a little bit, 2 = some what, 3 = quite a bit and 4 = very much, where the higher score indicated worse condition). Lymphoma subscale score is the total of reverse scores, range 0 to 60. Higher scores indicate a better quality of life.
Time Frame: Up to 8 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 28 | 28
months | 36.83 [4.86 to NA] — NA" represents that upper limit of 95% CI was not calculated due to insufficient number of participants with events. | 58.91 [5.82 to 85.88]

13. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. Adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE did not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs were defined as adverse events with onset or worsening on or after date of first dose of study treatment up to and including 30 days after date of last dose of study medication.
Time Frame: Placebo + Chemoimmunotherapy (CIT) arm: From Day 1 up to 30 days after date of last dose of study medication (up to 8 years); Ibrutinib + CIT arm: From Day 1 up to 30 days after date of last dose of study medication (up to 8 years 8 months)
Population: Safety analysis population included all randomized participants who received at least 1 dose of study drug, and were analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 199 | 201
Participants | 197 | 199

14. Secondary Outcome: Number of Participants With TEAEs: Participants With MZL
Description: Number of MZL participants with TEAEs were reported. AE was defined as any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE did not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs were defined as adverse events with onset or worsening on or after date of first dose of study treatment up to and including 30 days after date of last dose of study medication.
Time Frame: as for outcome 13
Population: Safety analysis population included all randomized participants with MZL who received at least 1 dose of study drug, and were analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
Number analyzed (Participants) | 28 | 28
Participants | 28 | 28

ADVERSE EVENTS:
Time Frame: All Serious AEs and Other (Not Including Serious) AEs: for Placebo + Chemoimmunotherapy (CIT) arm: From Day 1 up to 30 days after date of last dose of study medication (up to 8 years); Ibrutinib + CIT arm: From Day 1 up to 30 days after last dose of study medication (up to 8 years 8 months); all cause mortality: From Day 1 up to end of study (up to 9 years 1 month)
Description: All reported serious AEs and other AEs were analyzed on safety population: all randomized participants who received at least 1 dose of study drug, and were analyzed according to actual treatment received. All-cause mortality: ITT population - all randomized participants who were enrolled with FL/MZL and were analyzed according to treatment to which they were randomized. Placebo+CIT arm participants discontinued study treatment post primary analysis but were assessed for safety till end of study.
Arm/Group | Placebo + Chemoimmunotherapy (CIT) | Ibrutinib + CIT
All-Cause Mortality (participants affected / at risk) | 61/201 | 65/202
Serious Adverse Events (participants affected / at risk) | 76/199 | 113/201
Other Adverse Events (participants affected / at risk) | 196/199 | 198/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Chemoimmunotherapy (CIT) (N=199) | Ibrutinib + CIT (N=201)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 13
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 5
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 4
Cardiac Arrest (Cardiac disorders) | 2 | 0
Cardiac Dysfunction (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 3
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardiac Failure Chronic (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 2
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 2
Pericardial Effusion (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 | 1
Cataract Cortical (Eye disorders) | 0 | 1
Necrotising Retinitis (Eye disorders) | 0 | 1
Retinal Artery Occlusion (Eye disorders) | 1 | 0
Visual Impairment (Eye disorders) | 0 | 1
Abdominal Hernia (Gastrointestinal disorders) | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Anal Incontinence (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 1 | 1
Crohn's Disease (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenic Colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 2
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 1
Pharyngo-Oesophageal Diverticulum (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal Stenosis (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Chest Pain (General disorders) | 1 | 0
Gait Disturbance (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 0 | 2
Hernia (General disorders) | 0 | 1
Metaplasia (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Pelvic Mass (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 16
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0
Aspergillus Infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial Infection (Infections and infestations) | 0 | 1
Bacterial Sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 3
Campylobacter Gastroenteritis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 3 | 5
Chronic Sinusitis (Infections and infestations) | 0 | 1
Coronavirus Infection (Infections and infestations) | 0 | 1
Covid-19 Pneumonia (Infections and infestations) | 0 | 4
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus Chorioretinitis (Infections and infestations) | 1 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 2
Device Related Infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 2
Escherichia Pyelonephritis (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 1
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 2
Gingivitis (Infections and infestations) | 1 | 0
H1n1 Influenza (Infections and infestations) | 1 | 0
Haemophilus Infection (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Herpes Simplex (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 4 | 3
Infection (Infections and infestations) | 0 | 1
Infectious Pleural Effusion (Infections and infestations) | 0 | 1
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 0 | 1
Intervertebral Discitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 2
Nocardiosis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 2
Pelvic Abscess (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 9 | 20
Pneumonia Bacterial (Infections and infestations) | 0 | 2
Pneumonia Cytomegaloviral (Infections and infestations) | 1 | 1
Pneumonia Herpes Viral (Infections and infestations) | 0 | 1
Pneumonia Klebsiella (Infections and infestations) | 1 | 1
Pulpitis Dental (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 3 | 2
Rhinovirus Infection (Infections and infestations) | 0 | 2
Salmonella Sepsis (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 8
Septic Shock (Infections and infestations) | 1 | 3
Sinusitis (Infections and infestations) | 0 | 3
Skin Infection (Infections and infestations) | 0 | 1
Soft Tissue Infection (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 1 | 1
Staphylococcal Skin Infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3
Urinary Tract Infection (Infections and infestations) | 3 | 7
Urosepsis (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 0 | 1
Vascular Device Infection (Infections and infestations) | 0 | 1
Vestibular Neuronitis (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 1 | 0
Vulvitis (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 | 3
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 3
Platelet Count Decreased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypopharyngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Nasal Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of the Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 1
Post Herpetic Neuralgia (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Bipolar Disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Disinhibition (Psychiatric disorders) | 0 | 1
Psychiatric Decompensation (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 5
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Obstructive Nephropathy (Renal and urinary disorders) | 0 | 1
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Uterine Cyst (Reproductive system and breast disorders) | 0 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal Cord Leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Extremity Necrosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 2
Orthostatic Hypotension (Vascular disorders) | 2 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Chemoimmunotherapy (CIT) (N=199) | Ibrutinib + CIT (N=201)
Anaemia (Blood and lymphatic system disorders) | 39 | 50
Leukopenia (Blood and lymphatic system disorders) | 26 | 27
Lymphopenia (Blood and lymphatic system disorders) | 23 | 18
Neutropenia (Blood and lymphatic system disorders) | 69 | 75
Thrombocytopenia (Blood and lymphatic system disorders) | 28 | 46
Atrial Fibrillation (Cardiac disorders) | 5 | 12
Vertigo (Ear and labyrinth disorders) | 15 | 12
Abdominal Pain (Gastrointestinal disorders) | 18 | 16
Abdominal Pain Upper (Gastrointestinal disorders) | 13 | 19
Constipation (Gastrointestinal disorders) | 54 | 33
Diarrhoea (Gastrointestinal disorders) | 69 | 102
Dry Mouth (Gastrointestinal disorders) | 6 | 13
Dyspepsia (Gastrointestinal disorders) | 15 | 25
Nausea (Gastrointestinal disorders) | 78 | 103
Stomatitis (Gastrointestinal disorders) | 12 | 27
Vomiting (Gastrointestinal disorders) | 40 | 57
Asthenia (General disorders) | 16 | 16
Chills (General disorders) | 9 | 15
Fatigue (General disorders) | 60 | 73
Influenza Like Illness (General disorders) | 1 | 13
Malaise (General disorders) | 8 | 16
Oedema Peripheral (General disorders) | 18 | 18
Pyrexia (General disorders) | 45 | 60
Hypogammaglobulinaemia (Immune system disorders) | 7 | 20
Bronchitis (Infections and infestations) | 25 | 21
Cellulitis (Infections and infestations) | 2 | 16
Conjunctivitis (Infections and infestations) | 6 | 11
Covid-19 (Infections and infestations) | 4 | 15
Folliculitis (Infections and infestations) | 3 | 12
Gastroenteritis (Infections and infestations) | 11 | 10
Herpes Zoster (Infections and infestations) | 22 | 15
Influenza (Infections and infestations) | 16 | 17
Nasopharyngitis (Infections and infestations) | 31 | 23
Pneumonia (Infections and infestations) | 11 | 25
Respiratory Tract Infection (Infections and infestations) | 12 | 9
Sinusitis (Infections and infestations) | 12 | 15
Skin Infection (Infections and infestations) | 4 | 15
Upper Respiratory Tract Infection (Infections and infestations) | 49 | 47
Urinary Tract Infection (Infections and infestations) | 10 | 28
Fall (Injury, poisoning and procedural complications) | 3 | 12
Infusion Related Reaction (Injury, poisoning and procedural complications) | 18 | 15
Alanine Aminotransferase Increased (Investigations) | 23 | 27
Aspartate Aminotransferase Increased (Investigations) | 20 | 19
Blood Alkaline Phosphatase Increased (Investigations) | 3 | 15
Blood Bilirubin Increased (Investigations) | 13 | 9
Blood Creatinine Increased (Investigations) | 10 | 20
Lymphocyte Count Decreased (Investigations) | 14 | 17
Neutrophil Count Decreased (Investigations) | 27 | 32
Platelet Count Decreased (Investigations) | 17 | 35
Weight Decreased (Investigations) | 11 | 25
White Blood Cell Count Decreased (Investigations) | 29 | 31
Decreased Appetite (Metabolism and nutrition disorders) | 33 | 44
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 16
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 28
Back Pain (Musculoskeletal and connective tissue disorders) | 21 | 21
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 16 | 33
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 23
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 21 | 17
Dizziness Postural (Nervous system disorders) | 13 | 14
Dysgeusia (Nervous system disorders) | 3 | 12
Headache (Nervous system disorders) | 34 | 35
Neuropathy Peripheral (Nervous system disorders) | 10 | 12
Paraesthesia (Nervous system disorders) | 12 | 6
Peripheral Sensory Neuropathy (Nervous system disorders) | 8 | 12
Insomnia (Psychiatric disorders) | 16 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 57
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 16
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 20 | 18
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 11
Dry Skin (Skin and subcutaneous tissue disorders) | 9 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 25
Rash (Skin and subcutaneous tissue disorders) | 33 | 68
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 12 | 16
Hypertension (Vascular disorders) | 17 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/40/NCT01974440/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT01974440/SAP_001.pdf